CLINICAL TRIAL: NCT03872154
Title: Checklist-guided Shared Decision-making for Code Status Discussions in Medical Inpatients. A Cluster-randomized Multicenter Trial
Brief Title: Checklist-guided Shared Decision-making for Code Status Discussions in Medical Inpatients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Clinical Trial Unit, University Hospital Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Code status 2019
Record Dates: First submitted 2019-01-15; First posted 2019-03-13 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Code Status Discussions With Medical In-patients
Keywords: code status discussion; resuscitation; hospitalized patient; cardiac arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: cluster randomized
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): In this group (intervention), physicians will conduct checklist-guided shared decision making to determine the patient's code status. Additionally, physicians will be given a decision aid, which they are told to use to illustrate impact and outcome of in-hospital cardiac arrests.
  Ancillary project (patients considered as futile): In this group (intervention), physicians will conduct checklist-guided communication.
  Interventions: Other: Checklist-guided shared decision-making
- Usual Care (No Intervention): In this group (control), physicians will conduct code status discussions as usually.

INTERVENTIONS:
Other: Checklist-guided shared decision-making — Physicians will receive a checklist and a decision aid for shared decision-making during code status discussion.
  Ancillary project: Physicians will receive a checklist to communicate the futility.
  Arms: Intervention

SUMMARY:
This cluster-randomized, multicenter trial is designed to investigate the effect of checklist-guided shared decision-making including decision aids and communication of expected outcome on patients' decision regarding their code status, and at the same time, if it improves decision-making quality as judged by patient's decisional comfort, patient knowledge and involvement in decision-making and patient satisfaction. Patients in whom resuscitation is considered as futile will be treated separately in an ancillary project. In these patients a checklist to communicate the futility and the medical consequences will be used.

ELIGIBILITY:
Inclusion Criteria:

1. physician level

   - residents on the medical wards will be the primary level of randomization.
2. patient level - any adult (>18 years) patient that is admitted for in-hospital care will be eligible.

Exclusion Criteria:

1. physician level

   - no exclusion criteria for physicians except if they refuse participation
2. patient level

   * patients unable to complete questionnaires or unable to follow code status discussions due to (1) intoxication, (2) paracusis; (3) serious psychiatric conditions (e.g., psychosis, depression with suicidal tendency, stupor), (4) cognitive impairment (e.g. dementia, delirium).
   * patients prior included in this study (i.e., patients who are hospitalized for the second time)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2663 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Frequency of "Do Not Resuscitate" (DNR) code status | Within 24 hours after code status discussion which is performed once at baseline
  Frequency of patients that forego resuscitation measures in case of a cardiac arrest

SECONDARY OUTCOMES:
Key secondary endpoint: Decisional conflict assessed by Decisional conflict Scale | Within 24 hours after code status discussion
  Patients' comfort with decision assessed through a validated German translation of the Decisional conflict Scale (DCS) The DCS is a 16 item-scale grouped into five sub-scales: certainty, information, clarification of values, external support or pressure and the patients perception of the quality of the decision process The score ranges from 0 (no decisional conflict) to 100 (extremely high decisional conflict). According to literature, individuals whose scores are greater than 37.5 are uncomfortable with the decision and tend to delay it
Patients' involvement in shared decision-making process assessed by questionnaire | Within 24 hours after code status discussion
  Patients' involvement in shared decision-making (SDM) process assessed via a validated German translation of the SDM-q-9 questionnaire
  The SDM-q-9 is a 9-item instrument to measure the process of SDM in the medical consultation from the patients' perspective.
Patients' fears and concerns induced by code status discussion | Within 24 hours after code status discussion
  Patients' concerns brought up by the code status discussion e.g. general concerns, concern of suffering from a cardiac arrest, concern of being seriously ill, patient's perception of feeling under pressure to discuss code status, each rated on a visual analogue scale (VAS) 0-10
Patients' satisfaction with code status discussion and perceived quality | Within 24 hours after code status discussion
  Satisfaction with code status discussions and perceived quality e.g. satisfaction with discussion, perceived transparency of discussion, perceived comprehensibility of information, perceived right to be heard, how well questions were answered, perceived competence of resident, perceived resident's ability to listen to patient, each rated on a VAS 0-10
Patients' Knowledge | Within 24 hours after code status discussion
  Patient's Knowledge assessed by a Knowledge Assessment Questionnaire being used in previous studies This tool is a 6-item questionnaire with five true/false and one multiple choice question to assess patients understanding of resuscitation and medical care. Scores range from 0 to 6, with higher scores reflecting greater knowledge

CONTACTS AND LOCATIONS:
Overall Officials: Sabina Hunziker, Prof, Principal Investigator — University Hospial Basel
Locations (1):
- Universitätsspital Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Arpagaus A, Arpagaus L, Becker C, Gross S, Gossi F, Bissmann B, Zumbrunn SK, Schuetz P, Leuppi JD, Aujesky D, Hug B, Peters T, Bassetti S, Hunziker S. Checklist-Guided Code Status Discussions in Patients for Whom Cardiopulmonary Resuscitation Is Considered Futile: An Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2025 Sep 2;8(9):e2533638. doi: 10.1001/jamanetworkopen.2025.33638. PMID 40996760
- [Derived] Becker C, Gross S, Beck K, Amacher SA, Vincent A, Mueller J, Loretz N, Blatter R, Bohren C, Urben T, Arpagaus A, Schaefert R, Schuetz P, Kaegi-Braun N, Stalder L, Leuppi JD, Aujesky D, Baumgartner C, Hug B, Schmieg H, Delfine V, Peters T, Templeton AJ, Bassetti S, Hunziker S. A Randomized Trial of Shared Decision-Making in Code Status Discussions. NEJM Evid. 2025 May;4(5):EVIDoa2400422. doi: 10.1056/EVIDoa2400422. Epub 2025 Apr 22. PMID 40261118